CLINICAL TRIAL: NCT06164743
Title: A Phase 2, Double-masked, Randomized, Vehicle-controlled Study of VVN461 Ophthalmic Solution in Treating Post -Operative Ocular Inflammation in Subjects Undergoing Routine Unilateral Cataract Surgery
Brief Title: Phase 2: VVN461 Ophthalmic Solution for Post -Operative Ocular Inflammation After Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVN461-CS-201
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Double-masked, parallel, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked drug product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VVN461 1.0% (Experimental): VVN461 Ophthalmic Solution, 1.0%
  Interventions: Drug: VVN461 Ophthalmic Solution 1.0%
- VVN461 0.5% (Experimental): VVN461 Ophthalmic Solution, 0.5%
  Interventions: Drug: VVN461 Ophthalmic Solution 0.5%
- Vehicle (Placebo Comparator): VVN461 Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: VVN461 Ophthalmic Solution 1.0% — Topical ocular drug
  Arms: VVN461 1.0%
Drug: VVN461 Ophthalmic Solution 0.5% — Topical ocular drug
  Arms: VVN461 0.5%
Drug: Vehicle — Topical ocular drug
  Arms: Vehicle

SUMMARY:
This is a multicenter, double-masked, randomized, vehicle-controlled, parallel-comparison study conducted at sites in the United States (US) in subjects undergoing routine unilateral cataract extraction and lens replacement (CELR) surgery via phacoemulsification

DETAILED DESCRIPTION:
This is a phase 2, multicenter, double-masked, randomized, vehicle-controlled, parallel-comparison study conducted at sites in the US assessing the safety and ocular efficacy of VVN461 for treating post-operative ocular inflammation in subjects who undergo routine unilateral CELR surgery via phacoemulsification without surgical complication. Approximately 90 subjects (30 per group) will be randomized in a 1:1:1 ratio. Subjects will administer 1 eye drop in the study eye four times a day (QID) for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years of age and in good general health at Visit 1 (Screening)
* Willing and able to provide informed consent and provide relevant privacy authorization(s)
* Willing and able to comply with study requirements and visit schedule
* Clear ocular media (other than cataract) in the study eye
* Planning to undergo routine unilateral cataract surgery via phacoemulsification extraction and implantation of an intraocular lens.

Exclusion Criteria:

* Any ocular pain at Visit 1 (Screening)
* Recent use of corticosteroids or oral non-steroidal anti-inflammatory drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - United Medical Research Institute, Inglewood, California
  - North Bay Eye Associates, Petaluma, California
  - Martel Eye Associates, Rancho Cordova, California
  - ICON Eye Care, Grand Junction, Colorado
  - Levenson Eye Associates, Jacksonville, Florida
  - Comprehensive Eye Care, Ltd, Washington, Missouri
  - Center For Sight - Las Vegas, Las Vegas, Nevada
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Keystone Research, Austin, Texas
  - Houston Eye Associates, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VVN461 1.0% | VVN461 0.5% | Vehicle
Started | 30 | 30 | 31
Completed | 30 | 30 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VVN461 1.0% | VVN461 0.5% | Vehicle | Total
Number analyzed (Participants) | 30 | 30 | 31 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 7 | 25
  >=65 years | 21 | 21 | 24 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (7.28) | 68.5 (8.51) | 69.8 (7.94) | 69.1 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 18 | 55
  Male | 16 | 7 | 13 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 5 | 12
  White | 23 | 24 | 22 | 69
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 31 | 91

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell: Categorical Cure
Description: Proportion of subjects with grade of 0 using SUN Working Group Grading Scale (0 (none) to 4+ (>50 cells in field). Note - higher values represent a WORSE outcome.
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | VVN461 1.0% | VVN461 0.5% | Vehicle
Number analyzed (Participants) | 30 | 30 | 31
Participants | 18 | 16 | 6

2. Secondary Outcome: Safety of VVN461
Description: Number of subjects with Adverse Events
Time Frame: Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | VVN461 1.0% | VVN461 0.5% | Vehicle
Number analyzed (Participants) | 30 | 30 | 31
Participants | 2 | 3 | 3

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | VVN461 1.0% | VVN461 0.5% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT06164743/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT06164743/SAP_003.pdf